CLINICAL TRIAL: NCT01174381
Title: The Use of a Community-based Organization to Change Lifestyle Characteristics Related to Non Communicable Diseases: A Community Based Intervention Study Among 25-60 Year Olds
Brief Title: The Use of a Community-based Organization to Change Lifestyle Characteristics Related to Non Communicable Diseases
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Kelaniya (Other)
Responsible Party: Principal Investigator, T M E Dabrera, Doctor, University of Kelaniya
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: PGIM/AC/4
Record Dates: First submitted 2010-07-30; First posted 2010-08-03 (Estimated); Last update posted 2015-05-27 (Estimated); Status verified 2015-05

CONDITIONS: Diabetes; Hypertension; Stroke; Ischemic Heart Disease
Keywords: Non communicable disease; Lifestyle Modification; Community Based organization; community based study
MeSH Terms: conditions — Diabetes Mellitus; Hypertension; Stroke; Myocardial Ischemia; Noncommunicable Diseases

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Lifestyle modification (Experimental): Lifestyle modification for behavior change related to NCD prevention
  Interventions: Behavioral: lifestyle modification

INTERVENTIONS:
Behavioral: lifestyle modification — Lifestyle modification for six months

SUMMARY:
This study attempts to implement a lifestyle intervention programme aimed at changing the dietary habits, physical activity and alcohol and tobacco consumption in the 25-60year old adults in the MOH area, Ragama and measure the effectiveness of the programme.

DETAILED DESCRIPTION:
Sri Lanka as a developing nation needs to identify feasible and cost effective measures to face the epidemic of NonCommunicable Diseases(NCDs) in the future. Experiences gained over many years in the developed countries can be of great value in planning and implementing NCD prevention and control activities in the developing countries Results from many studies have emphasized the fact that merely providing risk reduction measures for clinically high-risk people in health service settings would have only a limited impact in the whole country. On the other hand, if the population as a whole were to be targeted, even a modest risk factor and healthy lifestyle change would potentially have a huge public impact.This study attempts to implement a lifestyle intervention programme aimed at changing the dietary habits, physical activity and alcohol and tobacco consumption in the 25-60year old adults in the MOH area, Ragama and measure the effectiveness of the programme. Outcome measures are process indicators, as measured by change in the dietary patterns, alcohol and tobacco consumption and physical activity. Short term outcome indicators would be blood pressure and anthropometric measurements. The long term outcome indicators such as morbidity and mortality due to NCD will not be measured as this will be a short term study.

ELIGIBILITY:
Inclusion Criteria:

* adults between 25-60 years

Exclusion Criteria:

* adults with psychiatric disorders

Ages: 25 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 440 (Actual)
Dates: Start 2010-08; Primary Completion 2011-01 (Actual); Study Completion 2011-02 (Actual)

PRIMARY OUTCOMES:
Proportion of participants who change their lifestyle characteristics related to NCDs | 6 months

SECONDARY OUTCOMES:
Proportion of participants with decrease in Body Mass Index following lifestyle modification programme | 6 months

CONTACTS AND LOCATIONS:
Overall Officials: Thushani M Dabrera, MBBS, MSc, Principal Investigator — University of Kelaniya
Locations (1):
- University of Kelaniya, Ragama, Western Province, Sri Lanka